CLINICAL TRIAL: NCT03611868
Title: A Phase Ib/II Study of APG-115 as a Monotherapy or in Combination With Pembrolizumab in Patients With Unresectable or Metastatic Melanomas or Advanced Solid Tumors
Brief Title: A Study of APG-115 in as a Monotherapy or Combination With Pembrolizumab in Patients With Metastatic Melanomas or Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG-115-US-002; Keynote B66 (Other: Merck and Co.); MK3475-B66 (Other: Merck and Co.)
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Unresectable or Metastatic Melanoma or Advanced Solid Tumors; Melanoma; Uveal Melanoma; P53 Mutation; MDM2 Gene Mutation; Cutaneous Melanoma; Mucosal Melanoma; Malignant Peripheral Nerve Sheath Tumors (MPNST)
Keywords: Metastatic melanoma, MPNST and Advanced Solid Tumors
MeSH Terms: conditions — Melanoma; Uveal Melanoma; Neurofibrosarcoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APG-115+pembrolizumab open label, two-part phase Ib/II (Experimental): single arm dose escalation and dose expansion
  Interventions: Drug: Phase 1b: APG-115+pembrolizumab

INTERVENTIONS:
Drug: Phase 1b: APG-115+pembrolizumab — dose escalation of APG-115 in combination with label dose of pembrolizumab, Four dose levels of APG-115 will be tested: 50, 100, 150, and 200 mg. APG-115 will be administrateddose escalation of APG-115 in combination with label dose of pembrolizumab, Fourfour dose levels of APG-115 will be tested: 50, 100, 150, and 200 mg. APG-115 will be administrated orally every other day (QOD) for consecutive 2 weeks (ie. dosed at Day 1, 3, 5, 7, 9, 11, and 13), with one week dosing off as there are cycles every 3-weeks a cycle. Pembrolizumab is administrated following FDA approved label dose, i.e., 200 mg intravenous infusion at Day 1 of every 3 weeks as a cycle.
  Phase II: Combination of APG-115 at 150 mg (RP2D) and pembrolizumab or APG-115 monotherapy alone.
  Other Names: KEYTRUDA®

SUMMARY:
This study aims to assess the safety, tolerability, pharmacokinetics, and preliminary efficacy of APG-115, an MDM2 inhibitor, either alone or in combination with pembrolizumab, a programmed cell death protein-1 (PD-1) inhibitor, in patients with metastatic melanomas or advanced solid tumors. Our hypothesis is that restoration of the immune response concomitant to inhibition of the MDM2 pathway (which restores p53 functions) may promote cancer cell death, leading to effective anticancer therapy.

DETAILED DESCRIPTION:
This is a phase I/II study to assess the safety and tolerability of APG-115 alone or in combination with pembrolizumab in patients with unresectable or metastatic melanoma, NSCLC, solid tumors with ATM mutation, liposarcoma, urothelial carcinomas, and malignant peripheral nerve sheath tumors (MPNST)The hypothesis is that the current therapy may improve ORR, progression-free survival, and synergistic effect of APG-115 alone or in combination with pembrolizumab in these patients. (n=230, ID: NCT03611868).

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female patients age ≥18 years, an exception for MPNST cohort: adolescents ≥12 years old (who weigh at least 40 kg) is allowed
* Part 2:

  1. Measurable disease according to RECIST 1.1. Lesions situated in a previously irradiated area, or an area subject to other loco-regional therapy (e.g., intralesional injections) should be considered non-measurable
  2. ECOG performance status 0-2
  3. Cohort A: Histologically confirmed, unresectable or metastatic melanoma, and refractory or relapse after PD-1 antibody treatment and ineligible for other standard of care therapy per NCCN guideline (previous PD-1/PD-L1 antibody treatment not required for uveal melanoma)
  4. Cohort F: Histologically confirmed, metastatic or unresectable MPNST
* Life expectancy ≥ 3 months
* Continuance of treatment related toxicities (except alopecia) due to prior radiotherapy or chemotherapy agents or biological therapy (including PD-1/PD-L1 antibodies) must be ≤ grade 1 at the time of dosing
* Adequate bone marrow and organ function without continuous supportive treatment
* QTcF interval (mean of 3, 1-3 minutes between tests) ≤450 ms in males and ≤470 ms in females
* Left ventricular ejection fraction (LVEF) ≥ lower limit of institutional normal (LLN) as assessed by echocardiogram (ECHO) or multigated acquisition (MUGA) scan
* Tumor tissue must be provided for all subjects for biomarker analysis before treatment with investigational product
* Willingness to use contraception by a method that is deemed effective by both male and female patients of childbearing potential and their partners throughout the treatment period and for at least three months following the last dose of study drug
* Ability to understand and willingness to sign a written informed consent form.

Exclusion Criteria:

* Any prior systemic MDM2-p53 inhibitor treatment
* Received chemotherapy within 21 days (42 days for nitrosoureas or mitomycin C) prior to first dose
* Part 2 Cohort A: Prior loco-regional treatment with intralesional therapy (e.g., talimogene laherparepvec) for unresectable or metastatic melanoma in the last 6 weeks prior to start of study treatment
* Part 2 Cohort B: Has received radiation therapy to the lung that is >30Gy within 6 months of the first dose of trial treatment
* Part 2 Cohort E: Known FGFR translocation mutation
* Received hormonal and biologic, small molecule targeted therapies or other anti-cancer therapy within 21 days prior to first dose
* Radiation or surgery within 14 days prior to first dose, thoracic radiation within 28 days prior to first dose
* Has known active central nervous (CNS) metastases and/or carcinomatous meningitis. Or has neurologic instability per clinical evaluation due to tumor involvement of the CNS.
* Requirement for corticosteroid treatment (with the exception of megestrol and local use of steroid: i.e., topical corticosteroids, inhaled corticosteroids for reactive airway disease, ophthalmic, intraarticular, and intranasal steroids
* Concurrent treatment with an investigational agent or device within 21 days prior to the first dose of therapy
* Failure to recover adequately, as judged by the investigator, from prior surgical procedures. Patients with active wound healing, patients who have had major surgery within 28 days from 1st dose of study treatment, and patients who have had minor surgery within 14 days from 1st dose of study treatment.
* Unstable angina, myocardial infarction, or a coronary revascularization procedure within 180 days of study entry
* Active rheumatoid arthritis (RA), active inflammatory bowel disease, chronic infections, or any other disease or condition associated with chronic inflammation
* Active infection requiring systemic antibiotic/ antifungal medication, and known clinically active viral infection such as hepatitis B or C, HIV infection, or active COVID-19
* Has received a live vaccine within 30 days prior to first dose.
* Has had an allogeneic tissue/solid organ transplant, prior stem cell or bone marrow transplant
* Has previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb)
* Any other condition or circumstance that would, in the opinion of the investigator, make the patient unsuitable for participation in the study
* History of organ transplant requiring use of immunosuppressive medication
* A woman of childbearing potential who has a positive urine or serum pregnancy test (within 72 hours) prior to treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2018-08-29 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 21 days
  Part I is to assess the safety and tolerability of APG-115 by assessing the dose-limiting toxicity (DLT) of APG-115 in combination with pembrolizumab. End points included: Incidence of DLTs during the first 3 weeks of treatment of each dose cohort; Severity and frequency of any adverse event(s) (AE) and serious adverse event(s) (SAE) based on NCI CTCAE 5.0
Recommended Phase II Dose | 21 days
  Part I is aimed to generate data to select the recommended Phase II dose
Overall Response Rate | up to 12 months
  Phase II is to assess overall response rate of APG-115 as monotherapy and in combination with pembrolizumab defined as the percentage of subjects with a best overall confirmed complete response (CR) or a partial response (PR) at any time as per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma
Locations (21):
- United States (17):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Highlands Oncology, Rogers, Arkansas
  - UCLA Hematology & Oncology Clinic, Los Angeles, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Children's National Research Institute, Washington D.C., District of Columbia
  - Sarah Cannon/FCSRI, Fort Myers, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Hershey Medical Center Cancer Institute, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Next Oncology, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Australia (4):
  - Metro South Hospital and Health Services via Princess Alexandra Hospital, Brisbane, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Austin Health, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: No